CLINICAL TRIAL: NCT05029206
Title: Hematopoietic Stem Cell Transplantation for Treatment of Multiple Sclerosis in Sweden - a Register-based Retrospective Observational Study
Brief Title: Hematopoietic Stem Cell Transplantation for Treatment of Multiple Sclerosis in Sweden
Acronym: AutoMS-Swe
Status: Completed | Type: Observational
Sponsor: Uppsala University (Other)
Collaborators: Karolinska University Hospital (Other); Sahlgrenska University Hospital (Other); Uppsala University Hospital (Other); Skane University Hospital (Other); University Hospital, Linkoeping (Other); University Hospital, Umeå (Other); Region Örebro County (Other)
Responsible Party: Sponsor
Other Study IDs: EPM 2021-01530
Record Dates: First submitted 2021-06-09; First posted 2021-08-31 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Multiple Sclerosis; Multiple Sclerosis, Relapsing-Remitting
Keywords: Autologous hematopoietic stem cell transplantation; Chemotherapy; Cyclophosphamide; Etoposide; Carmustine; Cytarabine; Melphalan; Antilymphocyte serum
MeSH Terms: conditions — Multiple Sclerosis; Multiple Sclerosis, Relapsing-Remitting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: Autologous hematopoietic stem cell transplantation — The therapeutic intervention of AHSCT consists of four parts: the mobilization of hematopoietic stem cells (HSC), the harvest of HSC, the ablation (conditioning) of the immune system and the reinfusion of autologous HSCs.
  1. In Sweden, the mobilization of HSCs has been made by a combination of cyclophosphamide (2 g/m2) and granulocyte-colony-stimulating factor.
  2. A minimum of 2 × 10^6 CD34+ cells/kg is harvested and cryopreserved. No in vitro manipulation is done to the stem cells.
  3. Two conditioning regimens have been used in Sweden for ablation. The BEAM-ATG protocol include carmustine (BCNU) 300 mg/m2, etoposide 800 mg/m2, cytarabine arabinoside (ARA-C) 800 mg/m2 and melphalan 140 mg/m2 + rATG or hATG. The Cy-ATG protocol include cyclophosphamide 200 mg/kg + rATG/hATG with 1000 mg Metylprednisolone given day -5 to -1.
  4. After a minimum of 24 hours after the last administration of chemotherapy have passed, the reinfusion of autologous CD34+ cells is performed.

SUMMARY:
This is an observational cohort study with retrospective analysis of prospectively collected data. The study cohort is constituted of all patients with relapsing-remitting multiple sclerosis (RRMS) treated with autologous stem cell transplantation (AHSCT) in Sweden from 2004 when the first AHSCT was performed until 31 December 2019. The study aims to describe the effectiveness, safety and patient reported outcomes of AHSCT for MS through real world data. Treatment related mortality will be analyzed from start of mobilization until the end of the study. For other adverse events the data collection will end 3 months post-transplantation. A statistical subgroup comparison of efficacy and safety between the conditioning regimens BEAM-ATG and Cy-ATG will be included within the study.

DETAILED DESCRIPTION:
All individuals with a diagnosis of MS, who was treated with AHSCT in Sweden until 31 December 2019 can be included in this study. Patients will be identified through the European Bone and Marrow Transplantation register (EBMT) and the Swedish MS register (SMSreg).

Baseline data will be collected from the SMSreg. Data concerning AHSCT will be collected from local repositories of the EBMT and supplemented by data obtained by reviewing of medical records. This includes data such as doses and names of drugs used for mobilization and conditioning, dates for administration of these drugs, date of hematopoietic stem cell transplantation, date of hematological milestones, occurrence and grading of adverse events during the first three months after the intervention.

Data on clinical outcome after the first three months of the intervention will be collected from SMSreg. Data on vital status will be collected from medical records at the end of study. Any recorded deaths will be analyzed through the medical records to determine if it was treatment-related.

The endpoints will be analysed and described for the whole study cohort. A subgroup analysis comparing the outcome of patients treated with different conditioning regimens (e.g. BEAM-ATG and Cy-ATG) will be included in this study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of multiple sclerosis according to the revised McDonald criteria 2017.
* Autologous hematopoietic stem cell transplantation performed for treating multiple sclerosis at a Swedish transplantation center until December 31st 2019.

Exclusion Criteria:

* Diagnosis of primary progressive MS or secondary progressive MS according to Lublin et al at the time of transplantation.
* Patient not accepted reporting of data to the EBMT register.
* Not fulfilling requirements of the minimal dataset, se below.

Definition of minimal dataset

* Data on disease course of multiple sclerosis at the time of transplantation.
* Transplantation and the following in-patient care performed in Sweden.
* Date of transplantation.
* Data on drugs used in conditioning.
* At least one follow-up visit performed in Sweden (unless early death before first follow-up visit) including data on:

  * Clinical assessment
  * The Kurtzke Expanded Disability Status Scores (EDSS)

Additional note: For a patient to be included in the analysis of treatment effectiveness data on MRI evaluation is needed at least once during follow-up.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All individuals with a diagnosis of MS, who was treated with AHSCT in Sweden until December 31st 2019 can be included in this study.
Sampling Method: Probability Sample
Enrollment: 174 (Actual)
Dates: Start 2021-05-05 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
No evidence of disease activity (NEDA) | 5 years
  NEDA is defined as absence of relapses in addition to absence of clinical progression and MRI progression.
Treatment related mortality (TRM) | Up to 18 years
  TRM is defined as death due to any transplantation-related cause other than disease progression.

SECONDARY OUTCOMES:
No evidence of disease activity (NEDA) | 3 years and 10 years
  NEDA is defined as absence of relapses in addition to absence of clinical progression and MRI progression.
MRI event free survival | At 3, 5 and 10 years
  The appearance of any T2 lesion > 3 mm or gadolinium enhancing lesion in the brain or spinal cord not present on the baseline scan measured from the time of AHSCT.
Relapse free survival | At 3, 5 and 10 years
  A clinical relapse defined as a period of acute worsening of neurological function lasting ≥ 24 hours not attributable to an external cause such as increased body temperature or acute infection, measured from the time of AHSCT.
Progression free survival | At 3, 5 and 10 years
  The Kurtzke Expanded Disability Status Scale (EDSS) is a method of quantifying disability in multiple sclerosis. The EDSS is a composite of disability in eight functional systems.
  Baseline EDSS ≤ 5 An increase in EDSS score with at least 1 point from baseline that is sustained between two follow-up visits separated in time by no less than six months.
  Baseline EDSS ≥ 5.5 An increase in EDSS score with at least 0.5 points from baseline that is sustained between two follow-up visits separated in time by no less than six months.
Annualized relapse rate (ARR) | Up to 17 years
  The number of relapses occurring during a time period divided by the number of years in that time period. E.g. 5 relapses occurring in a time period of 2.5 years equals an ARR of 2 (5/2.5=2), after AHSCT.
Proportion of patients with clinical improvement | Up to 17 years
  The Kurtzke Expanded Disability Status Scale (EDSS) is a method of quantifying disability in multiple sclerosis. The EDSS is a composite of disability in eight functional systems.
  Baseline EDSS ≤ 5.5 A decrease in EDSS score with at least 1 point from baseline that is sustained between two follow-up visits separated in time by no less than six months.
  Baseline EDSS ≥ 6 A decrease in EDSS score with at least 0.5 points from baseline that is sustained between two follow-up visits separated in time by no less than six months.
EDSS change | At 1, 2 and 3 years
  The Kurtzke Expanded Disability Status Scale (EDSS) is a method of quantifying disability in multiple sclerosis. The EDSS is a composite of disability in eight functional systems.
  Any change in EDSS from baseline to follow-up.
Grade 3 serious adverse events the first 100 days | 100 days
  The frequency and of grade 3 serious adverse events within 100 days as defined by the NIH common terminology criteria for adverse events (CTCAE).
Grade 4 serious adverse events the first 100 days | 100 days
  The frequency and of grade 3 serious adverse events within 100 days as defined by the NIH common terminology criteria for adverse events (CTCAE).

OTHER OUTCOMES:
Changes in cognitive function | At 1, 2 and 3 years
  Explorative outcome. Measured by Symbol Digit Modalities Test (SDMT) is a test of cognitive function in MS-patients.
Changes in quality of life | At 1, 2 and 3 years
  Explorative outcome. Changes in quality of life, measured by the Multiple Sclerosis Impact Scale (MSIS-29) from the patient's perspective.
Changes in MS-related fatigue | At 1, 2 and 3 years
  Explorative outcome. As measured by the Fatigue Scale for Motor and Cognitive Functions (FSMC), a 20-item scale for evaluating MS-related cognitive and motor fatigue.

CONTACTS AND LOCATIONS:
Overall Officials: Joachim Burman, MD, PhD, Principal Investigator — Uppsala University; Thomas Silfverberg, MD, Study Chair — Uppsala University
Locations (8):
- Sweden (8):
  - Sahlgrenska University Hospital, Gothenburg
  - Linköping University Hospital, Linköping
  - Skåne University Hospital, Lund
  - Örebro University Hospital, Örebro
  - Danderyd Hospital, Stockholm
  - Karolinska University Hospital, Stockholm
  - Umeå University Hospital, Umeå
  - Uppsala University Hospital, Uppsala

IPD SHARING:
Plan to Share IPD: Yes
Study protocol will be made available upon request.
Supporting Information: Study Protocol, CSR
Time Frame: The data set will be stored for 15 years
Access Criteria: Study protocol will be made available upon request. Access to study data will be decided after contact with the study principal investigator. All access should be of scientific purposes.

REFERENCES:
- [Background] Compston A, Coles A. Multiple sclerosis. Lancet. 2002 Apr 6;359(9313):1221-31. doi: 10.1016/S0140-6736(02)08220-X. PMID 11955556
- [Background] Bronnum-Hansen H, Koch-Henriksen N, Stenager E. Trends in survival and cause of death in Danish patients with multiple sclerosis. Brain. 2004 Apr;127(Pt 4):844-50. doi: 10.1093/brain/awh104. Epub 2004 Feb 11. PMID 14960501
- [Background] Daumer M, Griffith LM, Meister W, Nash RA, Wolinsky JS. Survival, and time to an advanced disease state or progression, of untreated patients with moderately severe multiple sclerosis in a multicenter observational database: relevance for design of a clinical trial for high dose immunosuppressive therapy with autologous hematopoietic stem cell transplantation. Mult Scler. 2006 Apr;12(2):174-9. doi: 10.1191/135248506ms1256oa. PMID 16629420
- [Background] Hader WJ. Disability and survival of multiple sclerosis in Saskatoon, Saskatchewan. Can J Neurol Sci. 2010 Jan;37(1):28-35. doi: 10.1017/s0317167100009616. PMID 20169770
- [Background] Skoog B, Runmarker B, Winblad S, Ekholm S, Andersen O. A representative cohort of patients with non-progressive multiple sclerosis at the age of normal life expectancy. Brain. 2012 Mar;135(Pt 3):900-11. doi: 10.1093/brain/awr336. PMID 22366800
- [Background] McFarland W, Granville NB, Dameshek W. Autologous bone marrow infusion as an adjunct in therapy of malignant disease. Blood. 1959;14(5):503-521. Blood. 2016 Apr 14;127(15):1839. doi: 10.1182/blood-2016-01-696450. PMID 27081092
- [Background] THOMAS ED, LOCHTE HL Jr, CANNON JH, SAHLER OD, FERREBEE JW. Supralethal whole body irradiation and isologous marrow transplantation in man. J Clin Invest. 1959 Oct;38(10 Pt 1-2):1709-16. doi: 10.1172/JCI103949. No abstract available. PMID 13837954
- [Background] Reiffers J, Trouette R, Marit G, Montastruc M, Faberes C, Cony-Makhoul P, David B, Bourdeau MJ, Bilhou-Nabera C, Lacombe F, et al. Autologous blood stem cell transplantation for chronic granulocytic leukaemia in transformation: a report of 47 cases. Br J Haematol. 1991 Mar;77(3):339-45. doi: 10.1111/j.1365-2141.1991.tb08581.x. PMID 1672819
- [Background] Philip T, Armitage JO, Spitzer G, Chauvin F, Jagannath S, Cahn JY, Colombat P, Goldstone AH, Gorin NC, Flesh M, et al. High-dose therapy and autologous bone marrow transplantation after failure of conventional chemotherapy in adults with intermediate-grade or high-grade non-Hodgkin's lymphoma. N Engl J Med. 1987 Jun 11;316(24):1493-8. doi: 10.1056/NEJM198706113162401. PMID 3295541
- [Background] Burt RK, Cohen BA, Russell E, Spero K, Joshi A, Oyama Y, Karpus WJ, Luo K, Jovanovic B, Traynor A, Karlin K, Stefoski D, Burns WH. Hematopoietic stem cell transplantation for progressive multiple sclerosis: failure of a total body irradiation-based conditioning regimen to prevent disease progression in patients with high disability scores. Blood. 2003 Oct 1;102(7):2373-8. doi: 10.1182/blood-2003-03-0877. Epub 2003 Jul 3. PMID 12842989
- [Background] Fagius J, Lundgren J, Oberg G. Early highly aggressive MS successfully treated by hematopoietic stem cell transplantation. Mult Scler. 2009 Feb;15(2):229-37. doi: 10.1177/1352458508096875. Epub 2008 Sep 19. PMID 18805841
- [Background] Burt RK, Loh Y, Cohen B, Stefoski D, Balabanov R, Katsamakis G, Oyama Y, Russell EJ, Stern J, Muraro P, Rose J, Testori A, Bucha J, Jovanovic B, Milanetti F, Storek J, Voltarelli JC, Burns WH. Autologous non-myeloablative haemopoietic stem cell transplantation in relapsing-remitting multiple sclerosis: a phase I/II study. Lancet Neurol. 2009 Mar;8(3):244-53. doi: 10.1016/S1474-4422(09)70017-1. Epub 2009 Jan 29. PMID 19186105
- [Background] Sormani MP, Muraro PA, Schiavetti I, Signori A, Laroni A, Saccardi R, Mancardi GL. Autologous hematopoietic stem cell transplantation in multiple sclerosis: A meta-analysis. Neurology. 2017 May 30;88(22):2115-2122. doi: 10.1212/WNL.0000000000003987. Epub 2017 Apr 28. PMID 28455383
- [Background] Sormani MP, Muraro PA, Saccardi R, Mancardi G. NEDA status in highly active MS can be more easily obtained with autologous hematopoietic stem cell transplantation than other drugs. Mult Scler. 2017 Feb;23(2):201-204. doi: 10.1177/1352458516645670. Epub 2016 Jul 11. PMID 27207454
- [Background] Rotstein DL, Healy BC, Malik MT, Chitnis T, Weiner HL. Evaluation of no evidence of disease activity in a 7-year longitudinal multiple sclerosis cohort. JAMA Neurol. 2015 Feb;72(2):152-8. doi: 10.1001/jamaneurol.2014.3537. PMID 25531931
- [Background] Burt RK, Balabanov R, Burman J, Sharrack B, Snowden JA, Oliveira MC, Fagius J, Rose J, Nelson F, Barreira AA, Carlson K, Han X, Moraes D, Morgan A, Quigley K, Yaung K, Buckley R, Alldredge C, Clendenan A, Calvario MA, Henry J, Jovanovic B, Helenowski IB. Effect of Nonmyeloablative Hematopoietic Stem Cell Transplantation vs Continued Disease-Modifying Therapy on Disease Progression in Patients With Relapsing-Remitting Multiple Sclerosis: A Randomized Clinical Trial. JAMA. 2019 Jan 15;321(2):165-174. doi: 10.1001/jama.2018.18743. PMID 30644983
- [Background] Muraro PA, Pasquini M, Atkins HL, Bowen JD, Farge D, Fassas A, Freedman MS, Georges GE, Gualandi F, Hamerschlak N, Havrdova E, Kimiskidis VK, Kozak T, Mancardi GL, Massacesi L, Moraes DA, Nash RA, Pavletic S, Ouyang J, Rovira M, Saiz A, Simoes B, Trneny M, Zhu L, Badoglio M, Zhong X, Sormani MP, Saccardi R; Multiple Sclerosis-Autologous Hematopoietic Stem Cell Transplantation (MS-AHSCT) Long-term Outcomes Study Group. Long-term Outcomes After Autologous Hematopoietic Stem Cell Transplantation for Multiple Sclerosis. JAMA Neurol. 2017 Apr 1;74(4):459-469. doi: 10.1001/jamaneurol.2016.5867. PMID 28241268
- [Background] Sharrack B, Saccardi R, Alexander T, Badoglio M, Burman J, Farge D, Greco R, Jessop H, Kazmi M, Kirgizov K, Labopin M, Mancardi G, Martin R, Moore J, Muraro PA, Rovira M, Sormani MP, Snowden JA; European Society for Blood and Marrow Transplantation (EBMT) Autoimmune Diseases Working Party (ADWP) and the Joint Accreditation Committee of the International Society for Cellular Therapy (ISCT) and EBMT (JACIE). Autologous haematopoietic stem cell transplantation and other cellular therapy in multiple sclerosis and immune-mediated neurological diseases: updated guidelines and recommendations from the EBMT Autoimmune Diseases Working Party (ADWP) and the Joint Accreditation Committee of EBMT and ISCT (JACIE). Bone Marrow Transplant. 2020 Feb;55(2):283-306. doi: 10.1038/s41409-019-0684-0. Epub 2019 Sep 26. PMID 31558790
- [Background] Atkins HL, Bowman M, Allan D, Anstee G, Arnold DL, Bar-Or A, Bence-Bruckler I, Birch P, Bredeson C, Chen J, Fergusson D, Halpenny M, Hamelin L, Huebsch L, Hutton B, Laneuville P, Lapierre Y, Lee H, Martin L, McDiarmid S, O'Connor P, Ramsay T, Sabloff M, Walker L, Freedman MS. Immunoablation and autologous haemopoietic stem-cell transplantation for aggressive multiple sclerosis: a multicentre single-group phase 2 trial. Lancet. 2016 Aug 6;388(10044):576-85. doi: 10.1016/S0140-6736(16)30169-6. Epub 2016 Jun 9. PMID 27291994
- [Background] Hamerschlak N, Rodrigues M, Moraes DA, Oliveira MC, Stracieri AB, Pieroni F, Barros GM, Madeira MI, Simoes BP, Barreira AA, Brum DG, Ribeiro AA, Kutner JM, Tylberi CP, Porto PP, Santana CL, Neto JZ, Barros JC, Paes AT, Burt RK, Oliveira EA, Mastropietro AP, Santos AC, Voltarelli JC. Brazilian experience with two conditioning regimens in patients with multiple sclerosis: BEAM/horse ATG and CY/rabbit ATG. Bone Marrow Transplant. 2010 Feb;45(2):239-48. doi: 10.1038/bmt.2009.127. Epub 2009 Jul 6. PMID 19584827
- [Background] Thompson AJ, Banwell BL, Barkhof F, Carroll WM, Coetzee T, Comi G, Correale J, Fazekas F, Filippi M, Freedman MS, Fujihara K, Galetta SL, Hartung HP, Kappos L, Lublin FD, Marrie RA, Miller AE, Miller DH, Montalban X, Mowry EM, Sorensen PS, Tintore M, Traboulsee AL, Trojano M, Uitdehaag BMJ, Vukusic S, Waubant E, Weinshenker BG, Reingold SC, Cohen JA. Diagnosis of multiple sclerosis: 2017 revisions of the McDonald criteria. Lancet Neurol. 2018 Feb;17(2):162-173. doi: 10.1016/S1474-4422(17)30470-2. Epub 2017 Dec 21. PMID 29275977
- [Background] Lublin FD, Reingold SC, Cohen JA, Cutter GR, Sorensen PS, Thompson AJ, Wolinsky JS, Balcer LJ, Banwell B, Barkhof F, Bebo B Jr, Calabresi PA, Clanet M, Comi G, Fox RJ, Freedman MS, Goodman AD, Inglese M, Kappos L, Kieseier BC, Lincoln JA, Lubetzki C, Miller AE, Montalban X, O'Connor PW, Petkau J, Pozzilli C, Rudick RA, Sormani MP, Stuve O, Waubant E, Polman CH. Defining the clinical course of multiple sclerosis: the 2013 revisions. Neurology. 2014 Jul 15;83(3):278-86. doi: 10.1212/WNL.0000000000000560. Epub 2014 May 28. PMID 24871874
- [Background] Alping P, Burman J, Lycke J, Frisell T, Piehl F. Safety of Alemtuzumab and Autologous Hematopoietic Stem Cell Transplantation Compared to Noninduction Therapies for Multiple Sclerosis. Neurology. 2021 Mar 16;96(11):e1574-e1584. doi: 10.1212/WNL.0000000000011545. Epub 2021 Jan 29. PMID 33514645
- [Background] Penner IK, Raselli C, Stocklin M, Opwis K, Kappos L, Calabrese P. The Fatigue Scale for Motor and Cognitive Functions (FSMC): validation of a new instrument to assess multiple sclerosis-related fatigue. Mult Scler. 2009 Dec;15(12):1509-17. doi: 10.1177/1352458509348519. Epub 2009 Dec 7. PMID 19995840
- [Background] Hobart J, Lamping D, Fitzpatrick R, Riazi A, Thompson A. The Multiple Sclerosis Impact Scale (MSIS-29): a new patient-based outcome measure. Brain. 2001 May;124(Pt 5):962-73. doi: 10.1093/brain/124.5.962. PMID 11335698
- [Background] Benedict RH, DeLuca J, Phillips G, LaRocca N, Hudson LD, Rudick R; Multiple Sclerosis Outcome Assessments Consortium. Validity of the Symbol Digit Modalities Test as a cognition performance outcome measure for multiple sclerosis. Mult Scler. 2017 Apr;23(5):721-733. doi: 10.1177/1352458517690821. Epub 2017 Feb 16. PMID 28206827